CLINICAL TRIAL: NCT06227559
Title: The Role of Some Hematological Parameters in Juvenile Systemic Lupus Erythematosus
Brief Title: The Role of Some Hematological Parameters in Juvenile Systemic Lupue Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Ali Mohamed Soliman Abdullah, Principal Investigator, Assiut University
Other Study IDs: Juvenile systemic lupus
Record Dates: First submitted 2023-12-17; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Juvenile systemic lupus erythematosus is an autoimmune disorder with multisystem involvement, leading to inflammatory damage to the joints, kidney, central nervous system, and hematopoietic system. Although the prevalence rate of juvenile systemic lupus erythematosus in a developing country is not known, as per literature the female-to-male ratio rises from 4.5 : 1 in adolescence to 8--12 : 1 in adult-onset patients.

- The full mechanism of SLE is still unknown however, production of autoantibodies and immune complex deposition with subsequent infiltration of neutrophils, hyper-activation of B and T cells, reduced ability of immune complexes and apoptotic cell clearance, and defects in multiple immune regulatory networks, are central to organ inflammation and subsequent damage in SLE. Systemic lupus erythematosus goes on with organ involvements by remission and relapses.

DETAILED DESCRIPTION:
Juvenile systemic lupus erythematosus is an autoimmune disorder with multisystem involvement, leading to inflammatory damage to the joints, kidney, central nervous system, and hematopoietic system. Although the prevalence rate of juvenile systemic lupus erythematosus in a developing country is not known, as per literature the female-to-male ratio rises from 4.5 : 1 in adolescence to 8--12 : 1 in adult-onset patients.

- The full mechanism of SLE is still unknown however, production of autoantibodies and immune complex deposition with subsequent infiltration of neutrophils, hyper-activation of B and T cells, reduced ability of immune complexes and apoptotic cell clearance, and defects in multiple immune regulatory networks, are central to organ inflammation and subsequent damage in SLE. Systemic lupus erythematosus goes on with organ involvements by remission and relapses.

The patients with SLE may present with various systemic manifestations. The general symptoms include: fever, malaise, arthralgias, myalgias, headache, and loss of appetite and weight. Nonspecific fatigue, fever, arthralgia, and weight changes.

- JSLE prognosis is related to the affected organs/systems and is worse for children and adolescents compared to adults, perhaps due to the higher rate of renal and neurological involvement attributed to JSLE.

Over the last decades, the improvement of patient survival was mainly due to an early diagnosis and better therapeutic approach, especially regarding the severe manifestations of the disease. These included the introduction of hemodialysis, renal transplantation and use of immunosuppressive drugs and their complications, i.e., use of potent antibiotic and hypertensive drugs .

* it is noteworthy that the hematological involvment predominates during the first years of the disease and tends to last over time, with the premise that it may be the initial manifestation of the disease. Clear examples of this are the cases of hemolytic anemia and immune thrombocytopenia that can be initially classified as idiopathic or primary to be later classified as secondary when associated with infections, medications, neoplasms, or autoimmune diseases. The spectrum of hematologic manifestations in SLE is very broad, including lymphopenia, anemia, thrombocytopenia, or pancytopenia.
* Platelet system activation is a key event in the pathogenesis of SLE. Circulating immune complexes, anti-phospholipid antibodies and infectious agents such as virus are the main activators of platelets in SLE. Neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) are two of the complete blood count parameters. A high NLR is used as an inflammatory marker for different autoimmune diseases. High PLR has been used as a marker for differential diagnosis or prognostic prediction of different diseases such as inflammatory diseases .

Over the past decade, PLR has emerged as a universal laboratory marker for predicting various neoplastic, prothrombotic, and metabolic diseases. PLR fluctuations can be interpreted in the context of the underlying multifaceted immune-inflammatory reactions. Shifts in this parameter correlate positively with other markers of systemic inflammation, particularly with NLR. PLR better predicts clinical outcomes in patients with systemic inflammation than either platelet or lymphocyte count .

* In previous studies, The major organ systems studied were: renal, hematological, cardiac, pulmonary, hepatic and the central nervous system. The results showed that a high percentage of children had hematological involvement (34%); thrombocytopenia (23%) and hemolytic anemia (20%).
* JSLE is not rare in Egypt and Africa, representing an important subset that is commonly over looked and requires special attention.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment ≤18 years old.
2. Both sexes
3. The Patients should be diagnosed as jSLE, according to 2019 European league against rheumatism (EULAR)/ American college of rheumatology (ACR) SLE classiﬁcation criteria, or the previous ACR 1997 SLE classification criteria.

Exclusion criteria:

1. Patients with autoimmune diseases other than j SLE
2. Patients not fulfilling the criteria for diagnosis of SLE
3. Active infections.
4. Malignancies.
5. Lymphoproliferative disorders.
6. Hematologic diseases
7. Hepatosplenic diseases and diabetic nephropathy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: this study will include all patients diagnosed and followed up as jSLE, and will be consecutively recruited from the inpatient and outpatient clinic of Immunology and rheumatology department at Assuit University children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Measure the absolute neutrophil-to-absolute lymphocyte ratio (NLR). | Baseline
  Measuring the absolute neutrophil-to-absolute lymphocyte ratio (NLR) by automated complete blood count ( 2 ml of venous blood will be obtained from the patients )
Measure the mean platelet volume (MPV). | Baseline
  Measuring the mean platelet volume (MPV) by automated complete blood count ( 2 ml of venous blood will be obtained from the patients )
Measure the platelet count-to-absolute lymphocytes ratio (PLR). | Baseline
  Measuring the platelet count-to-absolute lymphocytes ratio (PLR) by automated complete blood count ( 2 ml of venous blood will be obtained from the patients )
Measuring the monocyte distribution width (MDW)}. | Baseline
  Measuring the monocyte distribution width (MDW)} by automated complete blood count ( 2 ml of venous blood will be obtained from the patients )